CLINICAL TRIAL: NCT00556361
Title: Use of Ketamine Prior to Cardiopulmonary Bypass in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 28781 Bhutta; CUMG
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Ventricular Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Ventricular | interventions — Sodium Chloride; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: saline
- 2 (Experimental)
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: saline — 2 mg/Kg IV saline within 5 minutes of initiation of Cardiopulmonary bypass
  Arms: 1
Drug: ketamine — 2 mg/Kg IV within 5 minutes of cardiopulmonary bypass
  Arms: 2

SUMMARY:
To assess whether the drug ketamine given prior to cardiopulmonary bypass can decrease injury to the cells in the brain.

ELIGIBILITY:
Inclusion Criteria:

* less than one year of age
* undergoing cardiac surgery for repair of ventricular septal defect
* requiring cardiopulmonary bypass
* not requiring retrogrades cerebral perfusion

Exclusion Criteria:

* Downs Syndrome

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2004-07; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To compare expression of serum markers of CNS injury | within 48 hours
to compare expression of multiple pro and anti-inflammatory cytokines between cases and controls. | within 48 hours

SECONDARY OUTCOMES:
to compare the clinical, radiological and neurodevelopmental outcomes of the cases and controls | one month

CONTACTS AND LOCATIONS:
Overall Officials: Adnan T Bhutta, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Bhutta AT, Schmitz ML, Swearingen C, James LP, Wardbegnoche WL, Lindquist DM, Glasier CM, Tuzcu V, Prodhan P, Dyamenahalli U, Imamura M, Jaquiss RD, Anand KJ. Ketamine as a neuroprotective and anti-inflammatory agent in children undergoing surgery on cardiopulmonary bypass: a pilot randomized, double-blind, placebo-controlled trial. Pediatr Crit Care Med. 2012 May;13(3):328-37. doi: 10.1097/PCC.0b013e31822f18f9. PMID 21926656